CLINICAL TRIAL: NCT05600647
Title: Effectiveness of Magnetic Therapy With Exercise Versus Exercise Therapy in Old Patients With Chronic Mechanical Neck Pain
Brief Title: Magnetic Therapy Versus Exercise Therapy in Old Patients With Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Randa Mohammed Almasri, Principal investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGS-2020-03-082
Record Dates: First submitted 2022-06-05; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: Neck Pain; Magnetic therapy; Exercise; Elderly; Proprioception; Balance
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: the control group will receive the exercise program and the experimental group will receive the same exercise training program in addition to electromagnetic field therapy, three times per week for four weeks.
Who Masked: Outcomes Assessor
Masking Description: The assessment will be done by an independent assessor who will be blinded to the aim of the study and the patient's group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromagnetic Field therapy with an exercise program (Experimental): The magnetic field is generated through a mattress that is connected to the device. The maximum program, program 4, for 20 minutes with an intensity of 35 microtesla (level 10) and 50-60 Hz. Every patient is lying on the mattress in a supine position. In addition to exercise training program included postural correction strengthening exercises, stretching, proprioception and balance training
  Interventions: Device: Electromagnetic Field therapy with an exercise program
- exercise program (Active Comparator): Every patients will practice the exercise training program alone. the program included postural correction, strengthening exercises, stretching, proprioception and balance training
  Interventions: Other: exercise program

INTERVENTIONS:
Device: Electromagnetic Field therapy with an exercise program — 1. The magnetic field is generated through a mattress that is connected to the device. The maximum program, program 4, for 20 minutes with an intensity of 35 microtesla (level 10) and 50-60 Hz. the patient was lying on the mattress in a supine position.
  2. the exercise program included postural correction strengthening exercises, stretching, proprioception and balance training
  Other Names: BEMER 3000
  Arms: Electromagnetic Field therapy with an exercise program
Other: exercise program — the exercise program included postural correction, strengthening exercises, stretching, proprioception and balance training
  Arms: exercise program

SUMMARY:
Mechanical neck pain (MNP) is a common condition that affects all aging groups. MNP has a huge physical, psychological and economic impact. The aim of this study is to evaluate the effects of magnetic therapy (MT) with exercise versus exercise therapy on neck pain, proprioception, balance, and function in older patients with chronic MNP. Materials & Method: 50 male and female patients with chronic MNP, their ages will range from 56 years and above. They will be allocated from different physiotherapy departments. Eligible participants will be equally randomized into two groups. Group-I: 25 patients will practice the exercise training program in addition to receiving pulsed electromagnetic field therapy (PEMF) (experimental arm). Group-II: 25 patients will practice the exercise program.

All participants will receive three sessions every week for four weeks. The primary outcomes are pain (Visual Analogue Scale VAS) and balance (Single leg stance time test SLST, Tinetti balance assessment, and Timed Up and Go TUG). The secondary outcomes are the Neck Disability Index (NDI), cervical range of motion (CROM), cervical joint position sense error (JPSE), and quality of life QOL SF-36 questionnaire. Measurements will be taken before the first session, after two weeks, and after the last session.

DETAILED DESCRIPTION:
The aim of the study is to:

Evaluate effects of pulsed electromagnetic field therapy along with exercise versus exercise therapy alone on neck pain, proprioception, balance, QOL, and functions in elderly patients with chronic MNP.

Procedure Design of the study: Randomized clinical trial RCT. Subjects: 50 patients (male and female) will be recruited from two physiotherapy departments in Saudi Arabia according to the inclusion and exclusion criteria. Their age will be 56 and above years. The included participants will be equally randomized into one of two groups: Group-I: 25 patients will practice the exercise program in addition to receiving a pulsed electromagnetic field therapy (experimental arm). Group-II: 25 patients will practice the exercise program (control arm)_ Randomization is blocking randomization and will be taken by the main researcher using a random number generator by a computer program software http://mahmoodsaghaei.tripod.com/Softwares/randalloc.html#Generate. Allocation will be done by an independent person who is not involved in the study using concealed opaque envelopes.

Confidentiality: All participants' data will be saved in a personal computer locked with a password. All questionnaire papers will be kept with the primary researcher in a locker.

Patient's rights: All recruited patients will sign a consent form before their participation and they will be informed that the collected data might be published.

The recruited patients will be randomized into two groups:

Group-I: 25 male and female patients will practice the exercise program and PEMF using a Bio-Electro-Magnetic-Energy-Regulation (BEMER) device.

Group-II: 25 male and female patients will practice the exercise program. The BEMER has a weak, pulsed magnetic field. The magnetic field is generated through a mattress that is connected to the device. The device will be manually set on 50-60 Hz, intensity of 35 microtesla, for 20 minutes while the participant lying on the mattress in a supine position.

NB: Each patient in each group will receive three sessions per week for four weeks. Total number of sessions is 12 sessions. Received any newly prescribed pain medications such as anti-inflammatory or opioids will not be allowed for all participants to prevent their effects on the study results. The assessment will be repeated by the same blinded assessor after two weeks and after finishing the last session. All the measurements will be recorded in a table. In addition, the same assessment tools will be used for all patients in all the physiotherapy departments where the study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* chronic mechanical neck pain for > 3 months.
* pain at rest or with movement that is felt in the neck, shoulders, and between scapulas on VAS scale at least 3/10.
* did not have any physical therapy interventions in the last five weeks.

Exclusion Criteria:

* cognitive impairment, rheumatic disease, infected joints, uncontrolled cardiovascular or pulmonary diseases, neurological conditions or nerve pathology, radicular symptoms, or malignancy.
* previous cervical spine surgeries.
* implemented cardiac pacemakers or any other electrical devices.
* vestibular system dysfunction or internal ear problems.
* corticosteroid injection in the last 12 weeks before participation.
* lower limb pain or condition that prevents the participant from performing the standing balance assessment.

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 4 weeks
  Every patient was asked to but a mark on the VAS line which represents his/her level of neck pain intensity from 0 to 10.It is a 10 cm drawn line. Where 0 represents no pain and 10 is the maximum pain level. The patient will be asked to but a mark on the line which represents his/her level of pain.
Tinetti balance assessment | 4 weeks
  consists of 2 parts: balance (9 items) and gait (8 items) with a total score of 28. The test started with the patient sitting on armless chair then asked to stand up. The next step, then the assessor nudged the patient sternum to check the balance with the patient eyes opened and then closed then the patient turned around 360 degrees and lastly sat down. The next part was to test the gait to assess the dynamic balance. The patient had to walk about five meters on an even walkway in his usual walking pattern while the assessor assess the steps length, height, symmetry, and continuity and straightness of the trunk.
  24 is a low risk of falls, 19 to 23 is a moderate risk and 18 and less is a high risk of falls.
Single-leg stance time (SLST) | 4 weeks
  Every patient was asked to stand on the preferred leg for a maximum of 90 seconds with the arms on the sides. The elevated leg should not touch the other one. The test was performed with eyes opened first then repeated with eyes closed. The time was recorded with a stopwatch.with eyes open and closed will be used for static postural balance.The participant will stand on the preferred leg for a maximum of 90 seconds with the arms on the sides. The test will be performed with eyes opened first then with eyes closed. Time is recorded by a stopwatch.
Timed Up and Go | 4 weeks
  Every patient was asked to stand up from an armchair, walk for three meters (marked on the floor), and turn around the mark, go back and sit down again. Time was measured in seconds with a stopwatch.the patient will be asked to stand up from an armchair, walks for 3 meters (marked on the floor), and turns back and sits again. Time is measured in seconds with a stopwatch.

SECONDARY OUTCOMES:
Neck Disability Index | 4 weeks
  The scale consists of 10 items with six answers for each. These items are about reading, driving, lifting, personal care, hobbies and work activities, pain, concentration, sleep and headache. Scoring is from 0 to 100%, the higher the number the worse the disability.
Cervical range of motion (CROM) | 4 weeks
  It was measured using a goniometer device consisting of three inclinometers that are attached to a frame similar to eyeglasses. The rotation inclinometer needle is adjusted by a magnetic field which is produced by a black magnetic necklace. Measurements will be taken from a sitting position with eyes opened and without moving the upper trunk. The participant will be asked to move the neck actively into flexion, extension, lateral flexion, and rotation.
cervical joint position sense error test (JPSE) | 4 weeks
  It is used to measure cervical proprioception. It will be measured using the same ROM goniometer device but with the eyes closed. Every patient will be asked to try to relocate the head to a specific range, 50% of the active ROM, which is the target of the relocation of the neck. each direction will be repeated three times.
Quality of life questionnaire SF-36 | 4 weeks
  It was evaluated with Quality-of-life QOL SF-36. The higher the score the higher the satisfaction. it consists of 11 questions about the quality of life, function, social life, health, and psychological subscale. the higher the percentage the better the quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Imam abdulrahman bin faisal university, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The individuals date not shared but the final results comments will appear only